CLINICAL TRIAL: NCT01655303
Title: Oral Propranolol, Diltiazem, Metoprolol and Verapamil in Atrial Fibrillation Rate Control in Patients With Stable Hemodynamic Status
Brief Title: Rate Control in Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16057
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Rapid Ventricular Response Atrial Fibrillation
MeSH Terms: interventions — Propranolol; Metoprolol; Verapamil; Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- Metoprolol Per Oral (Experimental): 50 mg Metoprolol
  Interventions: Drug: Metoprolol
- Verapamil (Experimental): 40 mg Verapamil Per Oral
  Interventions: Drug: Verapamil
- Propranolol (Experimental): 40 mg Propranolol Per Oral
  Interventions: Drug: Propranolol
- Diltiazem (Experimental): 60 mg Diltiazem Per Oral
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Propranolol
  Other Names: Inderal
  Arms: Propranolol
Drug: Metoprolol
  Other Names: Metoral
  Arms: Metoprolol Per Oral
Drug: Verapamil
  Arms: Verapamil
Drug: Diltiazem
  Arms: Diltiazem

SUMMARY:
Rate control in atrial fibrillation is a usual battle in emergency departments. Oral medications have a natural superiority to intravenous ones because they are easy-to-use and decrease the workload in busy emergency departments.

This study wants to find an effective oral medication for rate control in rapid ventricular response atrial fibrillation. Propranolol and Metoprolol, Diltiazem and Verapamil are compared in patients with a stable hemodynamic status.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Stability in hemodynamic

Exclusion Criteria:

* Systolic blood pressure less than 90 mm Hg
* Altered mental status attributable to rapid ventricular response atrial fibrillation
* Acute pulmonary edema attributable to rapid ventricular response atrial fibrillation
* Chest pain attributable to rapid ventricular response atrial fibrillation
* Allergy to Propranolol or Metoprolol or Verapamil or Diltiazem
* History of asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rate less than 100 per minute | In 1 hour
  Ventricular rate less than 100 per minute after 1 hour of per oral medication administration

SECONDARY OUTCOMES:
Drugs adverse effects | 2 hours
  Drugs adverse effects seen in patients in 2 hours after per oral medication administration
Unstability in hemodynamic | 2 hours
  Hemodynamic instability (systolic blood pressure less than 90 mmHg, loss of consciousness, pulmonary edema, chest pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Rasoul-e-Akram Hospital, Tehran, Tehran Province, Iran